CLINICAL TRIAL: NCT04302675
Title: Adapting Motivational Interviewing for Maternal Immunizations (MI4MI)
Acronym: MI4MI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-1312; 1R21AI141822-01A1 (NIH)
Record Dates: First submitted 2020-02-25; First posted 2020-03-10 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Maternal Immunization
Keywords: Maternal Immunization; Immunization - Influenza; Immunization - Tdap; Tetanus; Diphtheria; Pertussis
MeSH Terms: conditions — Influenza, Human; Tetanus; Diphtheria; Whooping Cough

STUDY DESIGN:
Intervention Model Description: Pre-post feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention, Maternal Immunization (Experimental)
  Interventions: Behavioral: Prevention, Maternal Immunization

INTERVENTIONS:
Behavioral: Prevention, Maternal Immunization — This intervention will be focused on behavior change, both through providers gaining context, knowledge, confidence, and skills in talking to pregnant mothers about vaccination during pregnancy, but also with patients having increased knowledge about immunization issues, and decreased anxiety about getting vaccinated.
  There is only one intervention arm in this study, and this study is looking at prevention in a pre-post feasibility study.

SUMMARY:
Vaccinating pregnant women affords a unique opportunity to protect both mother and child against influenza and pertussis, yet uptake of maternal immunizations remain far below national target goals. A significant barrier to vaccine uptake is the lack of evidence to guide provider communication with patients who have concerns about vaccines. This novel study will adapt motivational interviewing to the ob-gyn setting to provide information about how to improve provider communication and increase vaccine uptake among pregnant women.

The investigators propose a pragmatic practice-based study in 5 ob-gyn practices in Colorado to develop the MI for maternal immunizations (MI4MI) intervention and assess fidelity, acceptability, and feasibility among patients and providers. Aim 1 will use an iterative process building upon existing knowledge of patient concerns about maternal immunizations and our prior experience training providers in Motivational Interviewing (MI) for childhood immunizations to develop the MI4MI training. During development, the study team will conduct focus groups to elicit provider input during. The MI4MI intervention will include a video-module, 2 asynchronous online trainings, provider reference sheets, and practice study champions. Aim 2 will include intervention implementation and assessment of intervention fidelity, acceptability, and feasibility. In Aim 2a, will conduct pre- and post-intervention chart reviews among participating practices to evaluate the impact of MI4MI on influenza and Tdap vaccine uptake among pregnant patients.

DETAILED DESCRIPTION:
Pertussis and influenza are the most poorly controlled vaccine preventable diseases in the United States. Pregnant women have increased risk of severe disease from influenza and newborns have increased risk of severe disease from influenza and pertussis. The Advisory Committee on Immunization Practices and American College of Obstetricians and Gynecologists recommend women receive influenza and pertussis (Tdap) vaccine during each pregnancy, yet only about half of pregnant women receive these vaccines. Among identified barriers to maternal immunization are patient concerns about vaccine safety and effectiveness and lack of evidence for how ob-gyn providers can best communicate vaccine recommendations. Interventions to address these barriers and increase uptake of maternal immunizations are urgently needed. Motivational interviewing (MI) is a communication technique that has proven effective for changing health behaviors including increasing adolescent vaccination rates. MI is both time-effective and acceptable to providers. The long-term goal of this project is to adapt MI to the ob-gyn setting to improve influenza and Tdap vaccine uptake in pregnancy. There is evidence to support use of MI for childhood immunizations; however it is unknown if MI is feasible and acceptable among ob-gyn providers and pregnant women. The investigators propose a pragmatic practice-based study in 5 Colorado ob-gyn practices to develop the MI for maternal immunizations (MI4MI) intervention and assess acceptability, adoption and implementation among patients and providers. Aim 1 will use an iterative process building upon existing knowledge of patient concerns about maternal immunizations and our prior experience training providers in MI for childhood immunizations to develop the MI4MI training. During development, the investigators will conduct focus groups for provider input and [organizational context. The MI4MI intervention will include a video-module, 2 asynchronous online trainings, provider reference sheets, and practice study champions. Aim 2 will include intervention implementation and assessment of MI4MI acceptability, adoption, and implementation. The study team will utilize patient "card study" surveys to assess the patient perspective of intervention acceptability. Patient surveys will be given to each pregnant patient seen for a prenatal visit during a 2-week period. We will interview up to 8 patient per practice after they fill out their card study to learn more about their interactions with providers and conversations around maternal immunizations. The investigators will conduct post-intervention provider focus groups to assess acceptability and adoption of the MI training intervention. The study team will also conduct pre-, interim-, and post-intervention surveys among providers to assess time spent and self-efficacy in vaccine communication. Providers will receive Maintenance of Certification or Continuing Medical Education credit for participation. In Aim 2a, investigators will conduct pre- and post-intervention chart reviews in study practices to evaluate the impact of MI4MI on influenza and Tdap vaccine uptake in pregnant patients. This study will provide data for a larger implementation study with rigorous assessment of the effectiveness of MI4MI in increasing maternal immunization uptake in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending ob-gyn practice in Colorado that is participating in the MI4MI project (5 total practices)
* Patients attending a pre-natal clinic visit at a participating practice during the intervention period who are eligible for maternal immunizations
* Pregnant patients who are less than 18 but 15 or more years of age will also be eligible to participate

Exclusion Criteria:

* Patients with hypersensitivity to any component of one of the recommended vaccines
* No subjects will be excluded because of ethnicity or insurance status.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participants must be currently pregnant, therefore anatomically female.
Enrollment: 1350 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
To develop the MI for maternal immunizations (MI4MI) provider training program | 12-18 months
  Based on the success of our MI program for vaccine hesitancy among parents of adolescents, we will use an iterative process [incorporating organizational perspectives and] provider feedback through focus groups to develop a multifaceted provider training program for using MI to encourage maternal immunization acceptance among women with concerns about vaccines. We will build upon existing knowledge of patient concerns to develop training in MI techniques with specific strategies to apply to maternal immunizations. The training intervention will include an online explainer video, two virtual interactive training modules, and provider reference sheets that can be used as an additional communication tool during the MI sessions with patients.

SECONDARY OUTCOMES:
To assess [acceptability, adoption and implementation] the MI4MI provider training program | 12-18 months
  We will conduct a pragmatic pilot study implementing the intervention in 5 Colorado ob-gyn practices. We will survey patients on their vaccine conversations with providers and interview up to 8 patients per practice to assess fidelity and adaptation of the intervention. These surveys will be conducted using a method known as a card study. Information gathered in the patient survey and subsequent interview will assess the acceptability of the intervention among patients who accept and refuse vaccines. We will conduct post-intervention focus groups among providers to assess the acceptability [and adoption] of the MI training intervention.
To evaluate the impact of the MI4MI intervention on vaccine acceptance among pregnant women | 12-18 months
  To assess [effectiveness], we will conduct chart reviews of study practices to compare Tdap and influenza vaccination rates in pregnant women pre- and post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sean O'Leary, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado at Denver and Health Sciences Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
No - We do not plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Brewer SE, Cataldi JR, Fisher M, Glasgow RE, Garrett K, O'Leary ST. Motivational Interviewing for Maternal Immunisation (MI4MI) study: a protocol for an implementation study of a clinician vaccine communication intervention for prenatal care settings. BMJ Open. 2020 Nov 17;10(11):e040226. doi: 10.1136/bmjopen-2020-040226. PMID 33203635

DOCUMENTS (1):
  • Informed Consent Form (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT04302675/ICF_000.pdf